CLINICAL TRIAL: NCT06267365
Title: Predictive Biomarker for Endoscopic Therapy in Chronic Pancreatitis
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23-00766
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (plasma/serum).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult Patients with Painful Chronic Pancreatitis: Participants with chronic pancreatitis scheduled for endoscopic therapy will undergo baseline assessments including EEG, quantitative sensory testing, and psychosocial questionnaires. Follow-up questionnaires will be completed at approximately 3, 6, 12 and 18 months post-procedure.

SUMMARY:
This is an observational prospective study to develop predictive biomarkers for pain response in participants with chronic pancreatitis scheduled for endoscopic therapy. Participants will undergo baseline assessments including electroencephalography (EEG), quantitative sensory testing (QST), and psychosocial questionnaires. Response to endoscopic therapy will be assessed at approximately 3, 6, 12 and 18 months post-procedure using questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* adults older than 18 years;
* Cambridge III or IV criteria for Chronic Pancreatitis (CP); or M-ANNHEIM criteria for definitive chronic pancreatitis;
* scheduled for endoscopic therapy for ductal obstruction (may include lithotripsy, pancreatic duct dilation, or stone extraction to facilitate successful stenting) as part of routine clinical care based on multidisciplinary review;
* pain present for ≥ 3 days per week for ≥ 3 months;
* average pain over the last week ≥ 4 on a 11-point numeric rating scale (NRS).

Exclusion Criteria:

* chronic pain syndrome other than CP;
* episode of acute pancreatitis within 2 months of enrollment;
* endoscopic therapy including Endoscopic retrograde cholangiopancreatography (ERCP), Endoscopic ultrasound (EUS) Guided Celiac Plexus Block or pancreatic surgery < 6 months prior to enrollment;
* active illicit drug use (excludes marijuana use);
* American Society of Anesthesiologists classification > 3;
* immune-mediated pancreatitis or associated pancreatic neoplasms
* Major neurological disease such as stroke, uncontrolled epilepsy, dementia
* Diagnosis of schizophrenia
* Chronic benzodiazepine use. Use of short acting benzodiazepine on as needed basis is acceptable if participant is able to hold benzodiazepine prior to EEG recording.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults older than 18 years with painful chronic pancreatitis scheduled for endoscopic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Brief Pain Inventory (BPI) Score at Month 3 Post-Operation | Baseline, Month 3 Post-Operation
  BPI is a 9-item assessment of pain. Each item is rated on a Likert scale from 0 (No Pain) to 10 (Pain as bad as you can imagine). The total score is the sum of responses and ranges from 0-90; higher scores indicate greater pain.

SECONDARY OUTCOMES:
Change from Baseline in BPI Score at Month 6 Post-Operation | Baseline, Month 6 Post-Operation
  BPI is a 9-item assessment of pain. Each item is rated on a Likert scale from 0 (No Pain) to 10 (Pain as bad as you can imagine). The total score is the sum of responses and ranges from 0-90; higher scores indicate greater pain.
Change from Baseline in BPI Score at Month 12 Post-Operation | Baseline, Month 12 Post-Operation
  BPI is a 9-item assessment of pain. Each item is rated on a Likert scale from 0 (No Pain) to 10 (Pain as bad as you can imagine). The total score is the sum of responses and ranges from 0-90; higher scores indicate greater pain.
Change from Baseline in BPI Score at Month 18 Post-Operation | Baseline, Month 18 Post-Operation
  BPI is a 9-item assessment of pain. Each item is rated on a Likert scale from 0 (No Pain) to 10 (Pain as bad as you can imagine). The total score is the sum of responses and ranges from 0-90; higher scores indicate greater pain.
Change from Baseline in Patient Reported Outcome System (PROMIS) - Physical Function - Short Form 6b Score at Month 3 Post-Operation | Baseline, Month 3 Post-Operation
  The PROMIS Physical Function Short Form 6b comprises 6 questions assessing general physical function. Each item is rated on a Likert scale from 1 (Unable to do) to 5 (Without any difficulty). The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater physical function.
Change from Baseline in PROMIS - Physical Function - Short Form 6b Score at Month 6 Post-Operation | Baseline, Month 6 Post-Operation
  The PROMIS Physical Function Short Form 6b comprises 6 questions assessing general physical function. Each item is rated on a Likert scale from 1 (Unable to do) to 5 (Without any difficulty). The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater physical function.
Change from Baseline in PROMIS - Physical Function - Short Form 6b Score at Month 12 Post-Operation | Baseline, Month 12 Post-Operation
  The PROMIS Physical Function Short Form 6b comprises 6 questions assessing general physical function. Each item is rated on a Likert scale from 1 (Unable to do) to 5 (Without any difficulty). The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater physical function.
Change from Baseline in PROMIS - Physical Function - Short Form 6b Score at Month 18 Post-Operation | Baseline, Month 18 Post-Operation
  The PROMIS Physical Function Short Form 6b comprises 6 questions assessing general physical function. Each item is rated on a Likert scale from 1 (Unable to do) to 5 (Without any difficulty). The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater physical function.
Number of Participants who use Opioids at Baseline | Baseline
Number of Participants who use Opioids at Month 3 | Month 3
Number of Participants who use Opioids at Month 6 | Month 6
Number of Participants who use Opioids at Month 12 | Month 12
Number of Participants who use Opioids at Month 18 | Month 18
Change from Baseline in PROMIS - Depression - Short Form 4a Score at Month 3 Post-Procedure | Baseline, Month 3 Post-Procedure
  The PROMIS Depression - Short Form 4a is a 4-item assessment of symptoms of depression in the past 7 days. Items are ranked on a Likert scale from 1 (never) to 5 (always). The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of depressive symptoms.
Change from Baseline in PROMIS - Depression - Short Form 4a Score at Month 6 Post-Procedure | Baseline, Month 6 Post-Procedure
  The PROMIS Depression - Short Form 4a is a 4-item assessment of symptoms of depression in the past 7 days. Items are ranked on a Likert scale from 1 (never) to 5 (always). The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of depressive symptoms.
Change from Baseline in PROMIS - Depression - Short Form 4a Score at Month 12 Post-Procedure | Baseline, Month 12 Post-Procedure
  The PROMIS Depression - Short Form 4a is a 4-item assessment of symptoms of depression in the past 7 days. Items are ranked on a Likert scale from 1 (never) to 5 (always). The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of depressive symptoms.
Change from Baseline in PROMIS - Depression - Short Form 4a Score at Month 18 Post-Procedure | Baseline, Month 18 Post-Procedure
  The PROMIS Depression - Short Form 4a is a 4-item assessment of symptoms of depression in the past 7 days. Items are ranked on a Likert scale from 1 (never) to 5 (always). The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of depressive symptoms.
Change from Baseline in PROMIS - Anxiety- Short Form 4a Score at Month 3 Post-Procedure | Baseline, Month 3 Post-Procedure
  The PROMIS Anxiety- Short Form 4a is a 4-item assessment of symptoms of anxiety in the past 7 days. Items are ranked on a Likert scale from 1 (never) to 5 (always). The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of anxiety.
Change from Baseline in PROMIS - Anxiety- Short Form 4a Score at Month 6 Post-Procedure | Baseline, Month 6 Post-Procedure
  The PROMIS Anxiety- Short Form 4a is a 4-item assessment of symptoms of anxiety in the past 7 days. Items are ranked on a Likert scale from 1 (never) to 5 (always). The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of anxiety.
Change from Baseline in PROMIS - Anxiety- Short Form 4a Score at Month 12 Post-Procedure | Baseline, Month 12 Post-Procedure
  The PROMIS Anxiety- Short Form 4a is a 4-item assessment of symptoms of anxiety in the past 7 days. Items are ranked on a Likert scale from 1 (never) to 5 (always). The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of anxiety.
Change from Baseline in PROMIS - Anxiety- Short Form 4a Score at Month 18 Post-Procedure | Baseline, Month 18 Post-Procedure
  The PROMIS Anxiety- Short Form 4a is a 4-item assessment of symptoms of anxiety in the past 7 days. Items are ranked on a Likert scale from 1 (never) to 5 (always). The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of anxiety.
Change from Baseline in PROMIS - Neuropathic Pain Quality 5a Score at Month 3 Post-Procedure | Baseline, Month 3 Post-Procedure
  The PROMIS Neuropathic Pain Quality 5a is a 5-item assessment of symptoms of neuropathic pain in the past 7 days. Items are ranked on a Likert scale from 1 (not at all) to 5 (very much). The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of neuropathic pain.
Change from Baseline in PROMIS - Neuropathic Pain Quality 5a Score at Month 6 Post-Procedure | Baseline, Month 6 Post-Procedure
  The PROMIS Neuropathic Pain Quality 5a is a 5-item assessment of symptoms of neuropathic pain in the past 7 days. Items are ranked on a Likert scale from 1 (not at all) to 5 (very much). The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of neuropathic pain.
Change from Baseline in PROMIS - Neuropathic Pain Quality 5a Score at Month 12 Post-Procedure | Baseline, Month 12 Post-Procedure
  The PROMIS Neuropathic Pain Quality 5a is a 5-item assessment of symptoms of neuropathic pain in the past 7 days. Items are ranked on a Likert scale from 1 (not at all) to 5 (very much). The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of neuropathic pain.
Change from Baseline in PROMIS - Neuropathic Pain Quality 5a Score at Month 18 Post-Procedure | Baseline, Month 18 Post-Procedure
  The PROMIS Neuropathic Pain Quality 5a is a 5-item assessment of symptoms of neuropathic pain in the past 7 days. Items are ranked on a Likert scale from 1 (not at all) to 5 (very much). The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of neuropathic pain.
Change from Baseline in PROMIS - Sleep Disturbance - Short Form 6a Score at Month 3 Post-Procedure | Baseline, Month 3 Post-Procedure
  The PROMIS Sleep Disturbance - Short Form 6a is a 6-item assessment of sleep disturbance in the past 7 days. Items are ranked on a Likert scale from 1-5. The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of sleep disturbance.
Change from Baseline in PROMIS - Sleep Disturbance - Short Form 6a Score at Month 6 Post-Procedure | Baseline, Month 6 Post-Procedure
  The PROMIS Sleep Disturbance - Short Form 6a is a 6-item assessment of sleep disturbance in the past 7 days. Items are ranked on a Likert scale from 1-5. The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of sleep disturbance.
Change from Baseline in PROMIS - Sleep Disturbance - Short Form 6a Score at Month 12 Post-Procedure | Baseline, Month 12 Post-Procedure
  The PROMIS Sleep Disturbance - Short Form 6a is a 6-item assessment of sleep disturbance in the past 7 days. Items are ranked on a Likert scale from 1-5. The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of sleep disturbance.
Change from Baseline in PROMIS - Sleep Disturbance - Short Form 6a Score at Month 18 Post-Procedure | Baseline, Month 18 Post-Procedure
  The PROMIS Sleep Disturbance - Short Form 6a is a 6-item assessment of sleep disturbance in the past 7 days. Items are ranked on a Likert scale from 1-5. The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of sleep disturbance.
Change from Baseline in PROMIS - Fatigue - Short Form 6a Score at Month 3 Post-Procedure | Baseline, Month 3 Post-Procedure
  The PROMIS Fatigue - Short Form 6a is a 6-item assessment of fatigue in the past 7 days. Items are ranked on a Likert scale from 1-5. The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of fatigue.
Change from Baseline in PROMIS - Fatigue - Short Form 6a Score at Month 6 Post-Procedure | Baseline, Month 6 Post-Procedure
  The PROMIS Fatigue - Short Form 6a is a 6-item assessment of fatigue in the past 7 days. Items are ranked on a Likert scale from 1-5. The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of fatigue.
Change from Baseline in PROMIS - Fatigue - Short Form 6a Score at Month 12 Post-Procedure | Baseline, Month 12 Post-Procedure
  The PROMIS Fatigue - Short Form 6a is a 6-item assessment of fatigue in the past 7 days. Items are ranked on a Likert scale from 1-5. The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of fatigue.
Change from Baseline in PROMIS - Fatigue - Short Form 6a Score at Month 18 Post-Procedure | Baseline, Month 18 Post-Procedure
  The PROMIS Fatigue - Short Form 6a is a 6-item assessment of fatigue in the past 7 days. Items are ranked on a Likert scale from 1-5. The raw score is the sum of responses and is transformed into a T-score a mean of 50 and standard deviation of 10. Scores range from 0-100; higher scores indicate greater prevalence of fatigue.
Change from Baseline in Pain Catastrophizing Scale (PCS) Score at Month 3 Post-Procedure | Baseline, Month 3 Post-Procedure
  The PCS is a 13-item assessment of the prevalence of thoughts and feelings associated with pain. Each item is rated on a Likert scale from 0 (not at all) to 4 (all the time). The total score is the sum of responses and ranges from 0 to 52; higher scores indicate greater pain catastrophizing.
Change from Baseline in PCS Score at Month 6 Post-Procedure | Baseline, Month 6 Post-Procedure
  The PCS is a 13-item assessment of the prevalence of thoughts and feelings associated with pain. Each item is rated on a Likert scale from 0 (not at all) to 4 (all the time). The total score is the sum of responses and ranges from 0 to 52; higher scores indicate greater pain catastrophizing.
Change from Baseline in PCS Score at Month 12 Post-Procedure | Baseline, Month 12 Post-Procedure
  The PCS is a 13-item assessment of the prevalence of thoughts and feelings associated with pain. Each item is rated on a Likert scale from 0 (not at all) to 4 (all the time). The total score is the sum of responses and ranges from 0 to 52; higher scores indicate greater pain catastrophizing.
Change from Baseline in PCS Score at Month 18 Post-Procedure | Baseline, Month 18 Post-Procedure
  The PCS is a 13-item assessment of the prevalence of thoughts and feelings associated with pain. Each item is rated on a Likert scale from 0 (not at all) to 4 (all the time). The total score is the sum of responses and ranges from 0 to 52; higher scores indicate greater pain catastrophizing.
Change from Baseline in Sleep Duration at Month 3 Post-Procedure | Baseline, Month 3 Post-Procedure
Change from Baseline in Sleep Duration at Month 6 Post-Procedure | Baseline, Month 6 Post-Procedure
Change from Baseline in Sleep Duration at Month 12 Post-Procedure | Baseline, Month 12 Post-Procedure
Change from Baseline in Sleep Duration at Month 18 Post-Procedure | Baseline, Month 18 Post-Procedure
Change from Baseline in Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Score at Month 3 Post-Procedure | Baseline, Month 3 Post-Procedure
  TAPS consists of a combined screening component (TAPS-1) followed by a brief followed by a brief assessment (TAPS-2) for those who screen positive. Scores on these questions generate a risk level per substance endorsed, based on a range of possible scores per substance. Scores range from 0-4; higher scores indicate a higher likelihood of problematic substance use.
Change from Baseline in TAPS Score at Month 6 Post-Procedure | Baseline, Month 6 Post-Procedure
  TAPS consists of a combined screening component (TAPS-1) followed by a brief followed by a brief assessment (TAPS-2) for those who screen positive. Scores on these questions generate a risk level per substance endorsed, based on a range of possible scores per substance. Scores range from 0-4; higher scores indicate a higher likelihood of problematic substance use.
Change from Baseline in TAPS Score at Month 12 Post-Procedure | Baseline, Month 12 Post-Procedure
  TAPS consists of a combined screening component (TAPS-1) followed by a brief followed by a brief assessment (TAPS-2) for those who screen positive. Scores on these questions generate a risk level per substance endorsed, based on a range of possible scores per substance. Scores range from 0-4; higher scores indicate a higher likelihood of problematic substance use.
Change from Baseline in TAPS Score at Month 18 Post-Procedure | Baseline, Month 18 Post-Procedure
  TAPS consists of a combined screening component (TAPS-1) followed by a brief followed by a brief assessment (TAPS-2) for those who screen positive. Scores on these questions generate a risk level per substance endorsed, based on a range of possible scores per substance. Scores range from 0-4; higher scores indicate a higher likelihood of problematic substance use.
Change from Baseline in Patient Global Impression of Change (PGIC) Score at Month 3 Post-Procedure | Baseline, Month 3 Post-Procedure
  PGIC is a 1-item assessment of patient's perception of the change in activity limitation, symptoms, emotions and overall quality of life related to their condition since beginning treatment. The item is rated on a scale from 1 (no change) to 7 (a great deal better). The final score is the numerical rating; higher scores indicate greater change.
Change from Baseline in PGIC Score at Month 6 Post-Procedure | Baseline, Month 6 Post-Procedure
  PGIC is a 1-item assessment of patient's perception of the change in activity limitation, symptoms, emotions and overall quality of life related to their condition since beginning treatment. The item is rated on a scale from 1 (no change) to 7 (a great deal better). The final score is the numerical rating; higher scores indicate greater change.
Change from Baseline in PGIC Score at Month 12 Post-Procedure | Baseline, Month 12 Post-Procedure
  PGIC is a 1-item assessment of patient's perception of the change in activity limitation, symptoms, emotions and overall quality of life related to their condition since beginning treatment. The item is rated on a scale from 1 (no change) to 7 (a great deal better). The final score is the numerical rating; higher scores indicate greater change.
Change from Baseline in PGIC Score at Month 18 Post-Procedure | Baseline, Month 18 Post-Procedure
  PGIC is a 1-item assessment of patient's perception of the change in activity limitation, symptoms, emotions and overall quality of life related to their condition since beginning treatment. The item is rated on a scale from 1 (no change) to 7 (a great deal better). The final score is the numerical rating; higher scores indicate greater change.
Change from Baseline in Patient Health Questionnaire-2 (PHQ-2) Score at Month 3 Post-Procedure | Baseline, Month 3 Post-Procedure
  PHQ-2 is a 2-item assessment of patient health in the last 2 weeks. Items are rated on a Likert scale from 0 (not at all) to 3 (nearly every day). The total score is the sum of responses and ranges from 0 to 6; lower scores indicate better health.
Change from Baseline in PHQ-2 Score at Month 6 Post-Procedure | Baseline, Month 6 Post-Procedure
  PHQ-2 is a 2-item assessment of patient health in the last 2 weeks. Items are rated on a Likert scale from 0 (not at all) to 3 (nearly every day). The total score is the sum of responses and ranges from 0 to 6; lower scores indicate better health.
Change from Baseline in PHQ-2 Score at Month 12 Post-Procedure | Baseline, Month 12 Post-Procedure
  PHQ-2 is a 2-item assessment of patient health in the last 2 weeks. Items are rated on a Likert scale from 0 (not at all) to 3 (nearly every day). The total score is the sum of responses and ranges from 0 to 6; lower scores indicate better health.
Change from Baseline in PHQ-2 Score at Month 18 Post-Procedure | Baseline, Month 18 Post-Procedure
  PHQ-2 is a 2-item assessment of patient health in the last 2 weeks. Items are rated on a Likert scale from 0 (not at all) to 3 (nearly every day). The total score is the sum of responses and ranges from 0 to 6; lower scores indicate better health.
Change from Baseline in Generalized Anxiety Disorder 2 (GAD-2) Score at Month 3 Post-Procedure | Baseline, Month 3 Post-Procedure
  GAD-2 is a 2-item assessment of symptoms of anxiety in the past two weeks. Items are rated on a Likert scale from 0 (not at all) to 3 (nearly every day).The total score is the sum of responses and ranges from 0-6; higher scores indicate greater symptoms of anxiety.
Change from Baseline in GAD-2 Score at Month 6 Post-Procedure | Baseline, Month 6 Post-Procedure
  GAD-2 is a 2-item assessment of symptoms of anxiety in the past two weeks. Items are rated on a Likert scale from 0 (not at all) to 3 (nearly every day).The total score is the sum of responses and ranges from 0-6; higher scores indicate greater symptoms of anxiety.
Change from Baseline in GAD-2 Score at Month 12 Post-Procedure | Baseline, Month 12 Post-Procedure
  GAD-2 is a 2-item assessment of symptoms of anxiety in the past two weeks. Items are rated on a Likert scale from 0 (not at all) to 3 (nearly every day).The total score is the sum of responses and ranges from 0-6; higher scores indicate greater symptoms of anxiety.
Change from Baseline in GAD-2 Score at Month 18 Post-Procedure | Baseline, Month 18 Post-Procedure
  GAD-2 is a 2-item assessment of symptoms of anxiety in the past two weeks. Items are rated on a Likert scale from 0 (not at all) to 3 (nearly every day).The total score is the sum of responses and ranges from 0-6; higher scores indicate greater symptoms of anxiety.
Change from Baseline in Pain, Enjoyment of Life and General Activity (PEG) Scale at Month 3 Post-Procedure | Baseline, Month 3 Post-Procedure
  PEG is a 3-item assessment of pain and how it interferes with activities of daily life. Each item is rated on a scale from 0 (does not interfere) to 10 (completely interferes). The total score is the average of the 3 items and ranges from 0-10; higher scores indicate greater pain interference.
Change from Baseline in PEG Scale at Month 6 Post-Procedure | Baseline, Month 6 Post-Procedure
  PEG is a 3-item assessment of pain and how it interferes with activities of daily life. Each item is rated on a scale from 0 (does not interfere) to 10 (completely interferes). The total score is the average of the 3 items and ranges from 0-10; higher scores indicate greater pain interference.
Change from Baseline in PEG Scale at Month 12 Post-Procedure | Baseline, Month 12 Post-Procedure
  PEG is a 3-item assessment of pain and how it interferes with activities of daily life. Each item is rated on a scale from 0 (does not interfere) to 10 (completely interferes). The total score is the average of the 3 items and ranges from 0-10; higher scores indicate greater pain interference.
Change from Baseline in PEG Scale at Month 18 Post-Procedure | Baseline, Month 18 Post-Procedure
  PEG is a 3-item assessment of pain and how it interferes with activities of daily life. Each item is rated on a scale from 0 (does not interfere) to 10 (completely interferes). The total score is the average of the 3 items and ranges from 0-10; higher scores indicate greater pain interference.

CONTACTS AND LOCATIONS:
Overall Officials: Tamas Gonda, MD, Principal Investigator — NYU Langone Health; Lisa Doan, MD, Principal Investigator — NYU Langone Health; Jing Wang, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
As an NIH-HEAL initiative sponsored study, our IPD sharing comply with the Helping to End Addiction Long-term (HEAL) Public Access and Data Sharing Policy. The de-identified participant data will be shared and deposited into the National Institute of Mental Health Data Archive (NIMH) Data Archive (NDA). The NDA provides metadata, study digital object identifier (DOI), and long-term access. This repository is supported by several institutes and centers at the NIH, and datasets are available through a request process. Investigators requesting data must be affiliated with an NIH-recognized research institution that maintains an active Federalwide Assurance (FWA), and complete and submit a Data Use Certification approved by an authorized institutional business official with signature authority. This request will then be reviewed by the NDA Data Access Committee.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Lisa.Doan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.